CLINICAL TRIAL: NCT05183659
Title: The Reliability of Myotonometer in Evaluating the Muscle Tone and Biomechanical Properties of the Forearm Muscles: Investigation of the Effect of Grip Strength on Mechanical Features
Brief Title: The Reliability of Myotonometer in Evaluating the Muscle Tone and Biomechanical Properties of the Forearm Muscles
Status: Completed | Type: Observational
Sponsor: İlke KARA, PT (Other)
Collaborators: Bitlis Eren University (Other); Dokuz Eylul University (Other)
Responsible Party: Sponsor-Investigator, İlke KARA, PT, Co-Principal Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Other Study IDs: BEU-IK-01
Record Dates: First submitted 2021-12-02; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Muscular Tone; Viscoelasticity
Keywords: elasticity; hardness; forearm muscles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study was to evaluate the intra-rater and inter-rater reliability of MyotonPRO in measuring muscle tone and mechanical properties of the wrist extensor and flexor muscles in healthy young adults. The secondary aim is to examine whether grip strength has any effect on muscle tone and biomechanical properties.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Body mass index < 30 kg/meter square
* Having no upper extremity injuries
* Willing and able to provide the written informed consent for the study

Exclusion Criteria:

* Use of medication that will affect muscle tone
* History of lateral or medial epicondylitis, trauma (elbow, hand or wrist), cervical radiculopathy, peripheral neuropathy or nerve injury (axillary, median, ulnar, radial, musculocutaneous), systemical diseases, muscle disorders (e.g. genetic diseases, neuromuscular disorders)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults between 18-35 years old
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Muscle tone (Hz) | Day 1
  The muscle tone which is a biomechanical property of the forearm muscles will be evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's biomechanical properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. To determine the feasibility of the MyotonPRO for assessing the muscle tone of forearm muscles measurements will be performed and recorded.
Stiffness (N/m) | Day 1
  The stiffness which is a biomechanical property of the forearm muscles will be evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's biomechanical properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. To determine the feasibility of the MyotonPRO for assessing the stiffness of forearm muscles measurements will be performed and recorded.
Elasticity (Logarithmic decrement) | Day 1
  The elasticity which is a viscoelastic property of the forearm muscles will be evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's viscoelastic properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. To determine the feasibility of the MyotonPRO for assessing the stiffness of forearm muscles measurements will be performed and recorded.

SECONDARY OUTCOMES:
Grip Strength | Day 1
  Handgrip strength will be measured with the JAMAR Hydraulic Hand Dynamometer. Participants will be asked to sit down with knees and hip flexed to 90⁰, forearm in a neutral position, wrist in 0-30⁰ extension, and 0-5⁰ ulnar deviation while on a chair with backrest. During the measurement, the examiner will instruct them to squeeze the handles of the dynamometer as strongly as possible and then let them loose completely, with a loud motivating command. This will be repeated 3 times with 1-minute rest breaks and the average value will be calculated. During the measurements, the Jamar dynamometer will be grasped from the lower and upper parts by the examiner.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No